CLINICAL TRIAL: NCT01385358
Title: A Study to Assess Catheter Ablation Versus Thoracoscopically Assisted Surgical Ablation in Persistent Atrial Fibrillation
Brief Title: Catheter Versus Thoracoscopic Surgical Ablation Strategy in Persistent Atrial Fibrillation
Acronym: CASA-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Wendy Butcher / Head of Research Governance and Performance, Royal Brompton & Harefield NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011CI004B; 11/SC/0032 (Other: Oxfordshire REC A Committee)
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracoscopically Assisted Surgical Ablation (Experimental): This arm will have an index thoracoscopically assisted surgical ablation.
  Interventions: Procedure: Thoracoscopically Assisted Surgical Ablation
- Catheter Ablation (Active Comparator): This is an active comparator arm where study subjects will undergo conventional catheter ablation.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Thoracoscopically Assisted Surgical Ablation — Surgical AF ablation including pulmonary vein isolation, gananglionated plexi ablation +/- LAA excision/exclusion.
  Arms: Thoracoscopically Assisted Surgical Ablation
Procedure: Catheter Ablation — In this arm, study subjects will undergo conventional catheter ablation as their index procedure. This will include pulmonary vein isolation, linear and electrogram based ablation.
  Arms: Catheter Ablation

SUMMARY:
Atrial fibrillation(AF)is the commonest arrhythmia worldwide and can lead to significant morbidity and mortality, posing an increasing public health burden. Restoration of sinus rhythm (SR) is the preferred strategy in symptomatic patients but outcomes with anti-arrhythmic drugs (AAD) are poor. The alternatives to AAD are two-fold.Firstly, catheter ablation (CA)- a technique that uses catheters (thin tubes) to deliver small 'heat lesions' to areas of the heart to eliminate AF. Secondly, surgical ablation, where multiple incisions are made in the atria to restore SR. Long term results from this traditional surgical approach are excellent however as it is technically difficult open-heart procedure with significant morbidity and mortality, it is seldom used.

CA is very effective in restoring SR in the early stages of AF when it is a paroxysmal (intermittent) rhythm disturbance. If not treated at this stage AF inevitably evolves into a more persistent or permanent state and becomes more difficult to treat with CA. Therefore, the optimum approach to treat patients with symptomatic long standing persistent AF has yet to be determined and remains a key area of on-going research.

New minimally invasive, thoracoscopically assisted surgical(closed-heart)approaches have recently developed which ablate a wide area around the pulmonary veins, and may offer advantages over the best current strategies in CA. There are also clear advantages for patients with greater safety and less discomfort when compared to traditional surgical open-heart procedures.

At present there is small amount of encouraging data on this thoracoscopic surgical technique but there is no data comparing these two modalities of treatment in persistent AF patients. The investigators therefore wish to prospectively investigate the safety and efficacy of this thoracoscopic surgical technique and compare with CA in this group of patients. MRI scanning will also be used to visualise the effects of ablation by analysis of scar formation.

The study hypothesises that thoracoscopics surgical ablation is a

DETAILED DESCRIPTION:
This will be a pilot, prospective, observational study of catheter ablation compared with thoracoscopically assisted, surgical ablation strategies using a case control design.

The study population will be patients between the ages of 18 and 80 with symptomatic long-standing persistent atrial fibrillation (≥1≤5 years) and good left ventricular function where at least one anti-arrhythmic drug (AAD) has failed, or where such drugs are contraindicated or not tolerated.

Thoracoscopically Assisted Surgical Ablation Group Patients assigned to this group will undergo minimally invasive, thoracoscopically assisted, surgical ablation to isolate the pulmonary veins (PVI) using a radiofrequency (RF) clamp device. This will include ganglionated plexi ablation +/- LAA excision/exclusion.

Catheter Ablation Group Patients will undergo pulmonary vein isolation, linear and electrogram based ablation.

Recurrences Only one redo procedure is allowed for atrial tachyarrhythmia recurrences in the 12 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 80
2. Symptomatic persistent AF (≥1≤5 years), refractory to at least 1 AAD and/or DCCV
3. Patient is legally competent and willing and able to sign informed consent form
4. Patient is willing and able to adhere to follow up visit protocols for the duration of the study

Exclusion Criteria:

1. Left ventricular ejection fraction < 40%
2. Cardiovascular implantable electronic device (contraindicates MRI imaging)
3. Contraindication to anticoagulation
4. Thrombus in the LA despite anticoagulation
5. CVA within the previous 6 months
6. Previous thoracic & cardiac surgery (including interventions for AF such as Cox-maze procedure)
7. Prior LA catheter ablation with the intention to treat AF
8. Prior AV nodal ablation
9. Patients actively participating in another research study will be not be permitted to enrol. Patients who have been involved with other research studies will be able to participate after a minimum period of 3 months after completion of prior study follow up.
10. Co-morbid condition that in opinion of investigator confers undue risk of GA or thoracoscopic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial tachyarrhythmias at 12 months. | 12 months
  Freedom from atrial tachyarrhythmias at 12 months which will be analysed with or without anti-arrhythmic drugs (AAD). Monitoring will be undertaken with ambulatory ECG monitoring in compliance with latest international guidelines.

SECONDARY OUTCOMES:
Freedom from atrial tachyarrhythmias at 12 months from a single procedure on/off AAD; | 12 months
  Only 1 re-do procedure is allowed in study time frame. But this outcome will look at single procedure success in both arms at 12 months.
Change in AF symptom score | Various time points 0,3,6,9,12 months
  Using recognised AF symptom score scale
Integrity of ablation lesion after index procedure at 3 months (as assessed by MRI if in SR +/- electrophysiologically if redo procedure is undertaken for atrial arrhythmia recurrence); | 3 months
  Using MRI +/- electrophysiological techniques.
Freedom of serious adverse events (stroke, myocardial infarction, emergency surgery, death) immediately after the procedure and during follow-up. | 12 months
Cost analysis (procedural and hospital stay costs). | 12 months
  Top down cost analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, Greater London, United Kingdom